CLINICAL TRIAL: NCT05995145
Title: A 8-week Randomized Controlled Trial of Active Mobilization of Hamstring for Non-specific Low Back Pain and Musculoskeletal Discomfort During Prolonged Sitting Among Young People: Study Protocol
Brief Title: Active Mobilization of Hamstring for Non-specific Low Back Pain and Musculoskeletal Discomfort During Prolonged Sitting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Józef Piłsudski University of Physical Education (Other)
Collaborators: University of Tehran (Other)
Responsible Party: Principal Investigator, Magdalena Plandowska, PhD, Józef Piłsudski University of Physical Education
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14/03/04/2023
Record Dates: First submitted 2023-07-29; First posted 2023-08-16 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2023-11

CONDITIONS: Low Back Pain
Keywords: exercise; treatment; spine; posture; students; pain; hamstring muscles
MeSH Terms: conditions — Low Back Pain; Motor Activity; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The hamstring stretching exercises program will be conducted five times a week, 20 min per session, for 8 weeks. The exercises will be supervised by an experienced physiotherapist with five years of clinical experience. The intervention will be divided into two parts. The first part will include exercises with a massage foam roller. The second part will include exercises of active hamstring flexibility exercises with hip flexion mobilization and the development of the habit of correct hip flexion technique, protecting the lower spine.
  Interventions: Behavioral: Active hamstring flexibility exercises with hip flexion mobilization
- Control group (No Intervention): Participants assigned to the control group will receive an self-care recommendations book.

INTERVENTIONS:
Behavioral: Active hamstring flexibility exercises with hip flexion mobilization — 8 weeks x 5 times per week for 20 min. In the experimental intervention, the exercise program will be based on participant education, home-based individual exercises, and regular group meetings for check-ups by a physiotherapist according to a precise set schedule.
  Arms: Experimental group

SUMMARY:
Hip flexion is a normal part of everyday functional activities, including walking and sitting. The length of the hamstring influences on movement of the pelvis during hip flexion, consequently influencing lumbar lordosis. In most activities, the hamstring muscles are active and it is necessary to keep them at normal length. Sitting posture is responsible for the loss of the natural curvature of the lumbar spine, because the hip flexion and pelvic extension flatten the lumbar vertebrae (i.e., lumbopelvic rhythm). Furthermore tightened hamstring increases posterior pelvic tilt and reduces lumbar lordosis, which can tend to low back pain (LBP). Stretching exercises play an important role in both the prevention and treatment of LBP. One important option will be exercise protocol which will combine the active hamstring flexibility exercises with hip flexion mobilization and the development of the habit of correct hip flexion technique, protecting the lower spine.

The aim of this RCT is to present a protocol for evaluating the effect of 8-week active hamstring flexibility exercises with hip flexion mobilization in reducing LBP and perceived musculoskeletal discomfort during prolonged sitting in young adults with non-specific LBP.

DETAILED DESCRIPTION:
Background:

Limited lower extremity muscle flexibility, such as hamstring, iliopsoas, quadriceps, and limited hip range of motion are risk factors for low back pain (LBP) in young people. LBP has increased by 49.8-50.7% over the last twenty years which highlighted the increase in the dominance of LBP especially among young people. Flexibility is an essential factor in physical fitness, which has a significant role in the functional development of the musculoskeletal system and the optimization of muscle work. To prevent pain or perceived musculoskeletal discomfort, various flexibility exercises including exercise stretches of the hamstring muscles have been recommended. Improving the hip flexion technique requires hip power and stability in the lumbar spine. In hamstring flexibility training, we should create an opportunity to practice movement and develop correct patterns using the hip flexion and extension pattern while maintaining the stability of the lumbar spine. Keeping the torso straight while working the hips and knees is one of the basic principles of protecting the spine in the lumbar region. Maintaining a neutral lower spine protects passive tissues and allows for better mobilization of the hips. Stretching exercises play an important role in both the prevention and treatment of LBP. One important option will be exercise protocol which will combine the active hamstring flexibility exercises with hip flexion mobilization and the development of the habit of correct hip flexion technique, protecting the lower spine.

Objective:

This randomized controlled trial aims to investigate the effect of a 8-week intervention involving active hamstring flexibility exercises with hip flexion mobilization on reducing low back pain (LBP) and perceived musculoskeletal discomfort during prolonged sitting in young adults with non-specific LBP.

Methods:

This will be a single-blind, randomized controlled trial with pre and post-intervention assessment. Participants were recruited from Physical Education Faculty students and randomly assigned to either the experimental group (hamstring stretching exercises) or the control group (no intervention). The hamstring stretching exercises group will be held five a week, 20 min per session for 8 weeks. The primary outcomes will be average pain intensity (Visual Analogue Scale, VAS), functional disability (Oswestry Disability Index), perceived musculoskeletal discomfort during prolonged sitting (Borg scale) , and the global perceived improvement (The Global Perceived Effect, 7-point Likert scale). Secondary outcome will be flexibility of the hamstring (SLR test).

Expected outcomes:

The findings of this study might provide information about a 8-week intervention involving active hamstring flexibility exercises with hip flexion mobilization on reduction of LBP and musculoskeletal discomfort during prolonged sitting in young adults. These results might highlight the importance of incorporating targeted flexibility exercises in the management of non-specific LBP, particularly in individuals with a sedentary lifestyle. Further research is warranted to explore the long-term effects and applicability of these interventions in larger populations.

ELIGIBILITY:
Inclusion Criteria:

* students in Physical Education (18-25 years old)
* with non-specific LBP (defined as pain and discomfort localized below the costal margin and above the inferior gluteal folds), the pain of at least 3 months duration, without radiation to legs
* without a surgical history due to spinal problems
* didn't previously continue the hamstring stretches exercises
* with hamstring muscle shortness

Exclusion Criteria:

* spinal pathology (eg, tumor, infection, fracture, inflammatory disease
* disc herniation and leg length discrepancy over 1cm
* pregnancy
* nerve root compromise
* previous spinal surgery
* major surgery scheduled during treatment or follow-up period
* presence of any contraindication to exercise
* medically verified chronic back disorde
* menstrual pain

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-02-12 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | Change from Pre-Intervention (baseline) compared to Post-Intervention (8 weeks)
  The Visual Analogue Scale (VAS) will be used to assess average pain intensity graded from 0 (no pain) up to 10 (unbearable pain). Mild pain or no pain will be defined as VAS 0-3, moderate pain as VAS 4-6, and severe pain as VAS 7-10. Participants will be asked to rate their maximum pain intensity from the last 3 months.
Functional Disability | Change from Pre-Intervention (baseline) compared to Post-Intervention (8 weeks)
  The Revised Oswestry Low Back Pain Disability Index will be used to assess the level of functional disabilities of participants resulting from LBP. The questionnaire consists of 10 items related to different aspects of function regarding activities of daily living (ADL). Each item will be scored from 0 to 5, with higher values representing greater disability. The total score will be multiplied by 2 and expressed as a percentage.
Perceived musculoskeletal discomfort during prolonged sitting | Change from Pre-Intervention (baseline) compared to Post-Intervention (8 weeks)
  The Borg CR-10 scale will be used to assess the perceived musculoskeletal discomfort during 1 hour of sitting named as prolonged sitting. The Borg CR-10 scale is presented in such a way that test subjects can indicate in which parts of the body feel discomfort (i.e. neck, shoulder, upper back, lower back, hip/thigh, and knee) and the degree of discomfort they feel (on a scale from 0 to 10, 0 being no discomfort and 10 being extremely uncomfortable).
The global perceived improvement | Completion of 8 week intervention
  The Global Perceived Effect (GPE) will be used to assess the global perceived improvement. The investigator will ask the student to rate, on a numerical scale, how much their condition has improved or deteriorated since some predefined time point: 1 = completely recovered, 2 = much improved, 3 = slightly improved, 4 = not changed, 5 = slightly worsened, 6 = much worsened and 7 = worse than ever. These ratings will be dichotomized into "improved" (GPE scores 1-2) and "not improved" (GPE scores 3 to 7).

SECONDARY OUTCOMES:
Flexibility of the hamstring | Change from Pre-Intervention (baseline) compared to Post-Intervention (8 weeks)
  The flexibility of the hamstring will be assessed through the SLR.The SLR is a passive test performed unilaterally. The criterion score of hamstring extensibility will be the maximum angle (degree) read from the goniometer at the point of maximum hip flexion. Angles will be recorded to the nearest degree for each leg. Two trials will give for each leg and the average of the two trials on each side will use for subsequent analysis. A subject's hamstring muscles will be considered tight (in a shortened position) if there was an SLR of ≤70 degrees.

CONTACTS AND LOCATIONS:
Locations (1):
- Jozef Pilsudski University of Physical Education in Warsaw, Faculty of Physical Education and Heath in Biala Podlaska, Biała Podlaska, Poland

IPD SHARING:
Plan to Share IPD: No